CLINICAL TRIAL: NCT01557179
Title: Evaluation of the Efficacy and Safety of Hyaluronic Acid Vaginal Gel to Ease Vaginal Dryness. A Multicenter, Randomized, Controlled, Open-label, Parallel-group, Clinical Trial
Brief Title: Evaluation of the Efficacy and Safety of Hyaluronic Acid Vaginal Gel to Ease Vaginal Dryness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEES_Hyalofemme_1; Hyalofemme (Registry Identifier: Hyalofemme)
Record Dates: First submitted 2012-03-14; First posted 2012-03-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: The Primary Objective of This Study Was to Assess the Efficacy and Safety of Hyaluronic Acid Vaginal Gel in Treating Vaginal Dryness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronic acid vaginal gel (Hyalofemme) (Experimental): The treatment in both groups was applied every 3 days for a total of 10 applications. Hyaluronic acid vaginal gel was supplied in a 30g aluminum tube with a vaginal applicator which provides a dose of around 5g
  Interventions: Device: Hyalofemme
- Estriol cream (Ovestin) (Active Comparator): The treatment in both groups was applied every 3 days for a total of 10 applications;Estriol cream was supplied in a 15g vial with a prefilled applicator providing a dose of around 0.5 g
  Interventions: Device: Estriol cream (Ovestin)

INTERVENTIONS:
Device: Hyalofemme — The treatment in both groups was applied every 3 days for a total of 10 applications. Hyaluronic acid vaginal gel was supplied in a 30g aluminum tube with a vaginal applicator which provides a dose of around 5g
  Arms: Hyaluronic acid vaginal gel (Hyalofemme)
Device: Estriol cream (Ovestin) — The treatment in both groups was applied every 3 days for a total of 10 applications;Estriol cream was supplied in a 15g vial with a prefilled applicator providing a dose of around 0.5 g
  Arms: Estriol cream (Ovestin)

SUMMARY:
This multicenter, randomized, controlled, open-label, parallel-group, 30-day study took place at four centers in China. The primary objective of this study was to assess the efficacy and safety of hyaluronic acid vaginal gel in treating vaginal dryness. In the current study we tested the hypothesis that the efficacy of hyaluronic acid vaginal gel was not inferior to that of estriol cream, with no clinically significant difference between them, in the treatment of vaginal dryness symptoms.

ELIGIBILITY:
Inclusion Criteria:

* under 70 years old,
* had been naturally or surgically postmenopausal for more than 6 months,
* had symptoms of vaginal dryness due to various causes and had no contraindications to locally applied estrogen

Exclusion Criteria:

* unmarried, pregnant and breast-feeding women,
* patients with vaginal infections such as trichomonas,
* candida and bacterial vaginosis,
* patients with breast cancer, uterine cancer or estrogen hormone dependent tumors,
* genital bleeding of unknown origin,
* patients with acute hepatopathy, embolic disorders,
* severe primary disease of the kidney and hematopoietic system
* recent malignant tumors

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
percentage of improvement of vaginal dryness symptoms | 30 days
  percentage of improvement of vaginal dryness symptoms at the baseline and after treatment

SECONDARY OUTCOMES:
percentage of improvement of itching, dyspareunia and burning sensation | 30 days
  percentage of improvement of itching, dyspareunia and burning sensation at baseline and after treatment